CLINICAL TRIAL: NCT01356771
Title: Melanoma Risk Assessment and Skin Cancer Awareness, Prevention, and Education in a Primary Care Setting
Brief Title: Melanoma Risk Assessment & Tailored Intervention
Acronym: PennSCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PennSCAPE; 5UC2CA148310-02 (NIH)
Record Dates: First submitted 2011-04-29; First posted 2011-05-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma; Skin Cancer
Keywords: Risk Assessment; Intervention
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Other)
  Interventions: Other: Surveys & Mailed Materials
- Tailored Intervention (Other): We will mail three separate pamphlets created specifically for the participant. The information in the pamphlets will be based on answers from the first survey.
  Interventions: Other: Surveys & Mailed Materials

INTERVENTIONS:
Other: Surveys & Mailed Materials — Phase I: Patients are screened for their level of risk for skin cancer. They will complete a survey and undergo a skin exam administered by the research staff. Moderate- and high-risk persons will be invited to enroll in Phase II.
  Phase II: Three sets of materials will be sent in the mail over the course of 6 weeks. Pamphlets will contain information about ways to reduce participant's risk of skin cancer, including sun protection practices, benefits of skin screening practices, and how to do skin self-examinations.
  The participant will also complete two surveys for this study, one at baseline and then one at follow up approximately three months later.
  Each survey will ask the participant about:
  * Current and past skin cancer screening practices
  * Current and past sun protection practices
  * Attitudes about skin cancer and sun protection
  * Knowledge of melanoma

SUMMARY:
The investigators are conducting a study to provide evidence about the comparative effectiveness of mailed, tailored intervention materials on cancer prevention behavioral outcomes. The investigators will send out three (3) tailored mailings for participants who are assigned to the intervention group. Second, during the eligibility screening, the investigators will be assessing the relative yield and functioning of two risk assessment tools (BRAT and FEARS) on determining an individual's level of risk for skin cancer.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of a mailed, tailored intervention, on the skin cancer prevention and skin self-examination behaviors of high-risk and moderate-risk adults. Participants will be recruited in primary health care setting (Penn Radnor Clinic) after their scheduled appointment. During Phase I of this study, patients will be screened for their level of risk for skin cancer. They will be asked to complete a survey as well as undergo a quick skin exam administered by the research staff. Moderate- and high-risk persons will be invited to enroll in Phase II of the study, and will then complete a baseline survey either in person, over the phone, or via mail after they have consented. After completing a baseline survey, these participants will be randomized to receive tailored materials, including personalized risk feedback, or to a control group that will receive generic educational materials. Participants will then be re-assessed at follow-up approximately three (3) months later via a mailed survey.

The intervention consists of one to three sets of intervention materials, depending on if they are randomized to the generic group or the tailored group. The first mailing will be sent out approximately two weeks after a participant completes the baseline survey, and is designed to educate participants on ways to prevent skin cancer though personalized behavioral changes. The second mailing will be sent out two weeks after the first mailing, and is designed to provide a guide to participants on steps to complete a skin self exam. Finally, the third mailing will be sent out two weeks after the second mailing, and will provide medical information to the participants regarding types of skin cancer along with tips to remember that encompass information from previous mailings.

Finally, the participant will complete a follow-up survey approximately one (1) month after the last mailing has been mailed.

ELIGIBILITY:
Inclusion Criteria:

To be included in Phase I, a subject must meet all of the following criteria:

1. Subjects are capable of giving informed consent
2. Subjects are ≥ 18 years old.
3. Subjects are English speaking and can read English

To be included for analysis during Phase II, a subject must meet all of the following criteria:

1. Subjects must meet all criteria listed in Phase I.
2. Subjects are identified as Caucasian.
3. Subjects must be at moderate or high risk for skin cancer, based on scores from the BRAT and Fears combined risk assessment.

Exclusion Criteria:

1. Children under the age of 18 will not be included.
2. For Phase II, previously diagnosed with melanoma.
3. For Phase II, planning to be away for three (3) consecutive weeks or longer in June, July, or August

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Compare the effects of offering tailored print materials to that of generic print materials on perceived risk of melanoma, sun avoidance/protection, and skin self-examination behaviors. | 3-6 months total per participant
  In Phase II of this study, we will conduct a randomized trial to compare the effects of a tailored intervention to a standard intervention of brochures with risk communication, skin cancer prevention, and skin cancer detection information. Outcomes are sun protection, sun exposure, frequency of sunburns, and skin examinations. Subjects in Phase II will be adults at moderate and high risk for skin cancer based on the scores they received from the risk assessment in Phase I.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Glanz, PhD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States